CLINICAL TRIAL: NCT01933893
Title: Follicular Versus Luteal Pipelle in Repeated Implantation Failure Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 139/13
Record Dates: First submitted 2013-08-29; First posted 2013-09-02 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Repeated Implantation Failure
Keywords: Pipelle, luteal, follicular, implantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
Pipelle was found to increase pregnancy and implantation rates in women undergoing IVF treatment in general, and in particular in repeated implantation failure (RIF). However, there is virtually no data regarding the optimal timing for the pipelle.

The current study aims to compare between follicular and luteal pipelle on pregnancy rate in RIF patients.

ELIGIBILITY:
Inclusion Criteria:

Women diagnosed with RIF who are going to start a new IVF treatment

Exclusion Criteria:

Known hydrosalpinx body mass index (BMI) >29 kg/m2 or <18 kg/m2 Low ovarian response

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women diagnosed with repeated implantation failure (RIF) who are undergoing IVF treatment.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | April, 2014

CONTACTS AND LOCATIONS:
Overall Officials: Ido Ben-Ami, MD, PhD, Principal Investigator — Assaf Harofeh Medical Center, Zerifin, Israel